CLINICAL TRIAL: NCT03484806
Title: China Registry and Cohort Study of Valvular Heart Disease in Adults
Brief Title: The China Valvular Heart Disease Study
Acronym: China-VHD
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yongjian Wu, coronary heart disease center, China National Center for Cardiovascular Diseases
Other Study IDs: 2017-I2M-3-002
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a observational、multicenter, prospective cohort study for adults with significant VHD. The purposes of this study were to evaluate the etiology、clinical characteristics、treatment modalities, and outcomes of patients with VHD；also to set up registration system of adult VHD in China, to build a database of Chinese adult VHD, to establish a web-based international standard data acquisition system for VHD and a multicenter clinical research platform. The results of the study will provide a basis for the future national health policy for prevention and treatment of adult VHD.

ELIGIBILITY:
Inclusion Criteria:

* patients over 60 years old meet one of the following conditions.

  1. moderate or above valvular heart disease as defined by echocardiography: （1）aortic stenosis, moderate or above, or valve area ≤1.5cm2, or maximal jet velocity ≥3.0m/sec, or mean pressure gradient ≥20mmHg, （2）aortic regurgitation, moderate or above, or jet width ≥25% of left ventricular outflow tract, or regurgitant volume ≥30ml/beat, or regurgitant fraction ≥30%, （3）mitral stenosis, moderate or above, or valve area ≤1.5cm2, （4）mitral regurgitation, moderate or above, or effective regurgitant orifice ≥0.2cm2, or regurgitant volume ≥30ml/beat, or regurgitant fraction ≥30%, （5）tricuspid stenosis, moderate or above, or valve area ≤1.0cm2, （6）tricuspid regurgitation, moderate or above, or central jet area ≥5.0cm2, （7）pulmonic stenosis, moderate or above, or maximal jet velocity >4m/sec, （8）pulmonic regurgitation, moderate or above,
  2. or patients who had undergone any operation on a cardiac valve (percutaneous balloon commissurotomy, valve repair, valve replacement, transcatheter aortic valve implantation),
  3. or diagnosis of endocarditis as assessed by Duke criteria.

Exclusion Criteria:

* Patients cannot be followed up for any reasons. Patients have been enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 60 years old with significant VHD
Sampling Method: Non-Probability Sample
Enrollment: 13917 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 2years

CONTACTS AND LOCATIONS:
Overall Officials: yongjian wu, doctor, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences; haiyan xu, doctor, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases，Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu X, Ye Y, Li Z, Liu Q, Zhao Z, Zhou Z, Wang W, Yu Z, Zhang H, Duan Z, Wang B, Zhang B, Lv J, Guo S, Zhao Y, Gao R, Xu H, Wu Y; China-VHD Study Collaborators. Primary regional disparities in clinical characteristics, treatments, and outcomes of a typically designed study of valvular heart disease at 46 tertiary hospitals in China: Insights from the China-VHD Study. Chin Med J (Engl). 2025 Apr 20;138(8):937-946. doi: 10.1097/CM9.0000000000003570. Epub 2025 Mar 18. PMID 40097371
- [Derived] Zhao Q, Zhang B, Ye Y, Li Z, Liu Q, Zhao R, Zhao Z, Wang W, Yu Z, Zhang H, Duan Z, Wang B, Lv J, Guo S, Zhao Y, Gao R, Xu H, Wu Y. Prognostic Impact of Left Ventricular Ejection Fraction in Patients With Moderate Aortic Regurgitation: Potential Implications for Treatment Decision-Making. Front Cardiovasc Med. 2022 Jan 17;8:800961. doi: 10.3389/fcvm.2021.800961. eCollection 2021. PMID 35111828